CLINICAL TRIAL: NCT06738940
Title: Long-term CPAP Effect on Social Jet Lag, Intake, Muscular Lipid, Hormone, and Cognition in Patients with Obstructive Sleep Apnea: a Telemedicine-based, Multi-center, Randomized Controlled Trial
Brief Title: Long-term CPAP Effect with Obstructive Sleep Apnea: a Telemedicine-based
Acronym: MSLS-LT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202402098DINC
Record Dates: First submitted 2024-11-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Body composition; Continuous positive airway pressure; Obstructive sleep apnea; social jet lag; cognition; muscular lipid
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use of CPAP device (Experimental): CPAP 48 weeks
  Interventions: Device: CPAP
- Usual care (No Intervention): Usual care 48 weeks

INTERVENTIONS:
Device: CPAP — Auto-CPAP treatment (AirSense™ 10 Autoset™, ResMed Inc., Australia) for 48 weeks
  Arms: Use of CPAP device

SUMMARY:
we hypothesize that long-term CPAP could results in increase weight and muscle composite by changing intake content and hormone and the effect was influenced by presence of CVD, social jet lag, and CPAP compliance. The project aims to conduct a telemedicine-based, multicenter, RCTs to compare the effect of 48-week CPAP and usual care on social jet lag, muscular fat, hormone, and attention and memory in 100 participants with moderate-severe OSA.

DETAILED DESCRIPTION:
After the participants enter the trial, participants underwent two-night home PSG to confirm the diagnosis of OSA. Once AHI ³15/h is confirmed, participants undertake baseline evaluation within two weeks which included standard questionnaire, eating behavior, 3-day photograph-based intake recording, and 7-day sleep log, 24-hr ambulatory blood pressure, 7-day Actiwatch and Actigraph, 2-morning attention and memory task at home environment. The BMR, BC, Proton Magnetic Resonance Spectroscopy (1H-MRS), and blood sampling are conducted in the morning when patients was fasting at hospital.

Once participants complete the baseline evaluation, they are randomly allocated to the usual care or auto-CPAP treatment (AirSense™ 10 Autoset™, ResMed Inc., Australia) for 48 weeks. The randomization is generated by the staff of the Department of Biostatistics independent of subject enrolment. A block-randomized assignment with a block size of four is used. Consecutive patients are assigned to the allocation according to the randomization schedule by the study nurse.

After randomization, participants had virtual visits at 4th, 12th, 24th, and 48th week and are evaluated with the same measurements as pre-randomization after complete the trial.

Once the patients complete the trial, they receive the standard treatment of OSA and are followed every 24 to 48 weeks for five years.

ELIGIBILITY:
Inclusion Criteria:

1. age:≧20 year-old
2. patients with moderate-severe OSA (AHI≥15/hr)

Exclusion Criteria:

1. skin allergy
2. wrist tattoos
3. BMI≧40 kg/m2
4. Neurological Disorders(Infection, Stroke, ALS, Myopathy, Brain tumor and Encephalitis)
5. Internal Diseases(cardiovascular disease or coronary artery disease was poorly controlled
6. chronic heart failure(including NYHA class 3 or more than NYHA class 3)
7. COPD(FEV1/FVC<70)
8. Hyperthyroidism or Hypothyroidism
9. Primary Aldosteronism
10. Chronic Kidney Disease(eGFR<30)
11. Acromegaly and Parkinson's disease)
12. Psychosis(Schizophrenia, bipolar disorder and depression)
13. Autoimmune disease(System Lupus Erythematosus, Rheumatoid arthritis, Sarcoidosis, Crohn's disease and Ulcerative Colitis)
14. Cancer(in last 5 years)
15. Have been diagnosed with obstructive sleep apnea
16. other sleep disorder(Narcolepsy, insomnia and RBD)
17. Use anti-inflammatory drugs(in last 2 weeks)
18. Illiterate
19. shift worker
20. has been Spinal Surgery and move difficult
21. professional driver has severe drowsiness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI | 12 months
  By comparing the BMI of the CPAP group and the usual care group, observe the effect of CPAP on BMI.
Changes in fat free mass | 12 months
  By comparing the fat free mass of the CPAP group and the usual care group, observe the effect of CPAP on fat free mass. Fat free mass was measured via bioelectrical impedance analysis (X-SCAN PLUS II, Jawon Medical Co., Ltd., Korea).

SECONDARY OUTCOMES:
The difference before and after the treatment of mid-sleep time | 12 months
  Evaluate mid-sleep time using the Actiwatch (Spectrum Plus, Philips Respironics, USA) and compare the differences between the CPAP group and the Usual Care group.
The difference before and after the treatment of BMR (REE) | 12 months
  The difference in BMR(Basal metabolic rate) between the CPAP group and the usual care group. The comparison item is REE(Resting Energy Expenditure) (kcal/day)
The difference before and after the treatment of BMR (RQ) | 12 months
  The difference in BMR(Basal metabolic rate) between the CPAP group and the usual care group. The comparison item is RQ(Respiratory Quotient) (kcal/day). The calculation method for RQ is to divide the amount of carbon dioxide (CO2) exhaled during BMR by the amount of oxygen (O2) consumed.
The difference before and after the treatment of Participants' nutrition intake | 12 months
  Energy intake was recorded via food diaries and photographs of intake for 3 days. Compare the differences between the CPAP group and the usual care group.
The difference before and after the treatment of attention and memory task | 12 months
  attention and memory task from E-Prime 3.0 software (Psychology Software Tools, Pittsburgh, PA, USA). Compare the differences between the CPAP group and the usual care group.

OTHER OUTCOMES:
Evaluate the difference between the usual care group and the CPAP group by comparing the activity levels measured by the Actiwatch and the sleeplog filled out by the patients. | 12 months
  After wearing the Actiwatch(Spectrum Plus, Philips Respironics, USA) for 7 days and recording the sleep log for 7 days, the bedtime and wake-up time recorded by the device will be compared with the bedtime and wake-up time reported by the patient to identify any discrepancies. This will be used to compare the pre- and post-treatment differences between the usual care group and the CPAP group.
The difference before and after the treatment of Biochemistry, hormone and cytokine(blood test) | 12 months
  Through CPAP treatment, blood test results for cortisol, lipid profile (T-CHO, TG, LDL, HDL), hsCRP, glucose, and insulin are expected to show differences in levels compared to pre-treatment values. This will be used to compare the usual care group and the CPAP group, in order to demonstrate the effectiveness of CPAP treatment.
The difference before and after the treatment of 24h blood pressure | 12 months
  The difference in 24-h systolic, diastolic(mmHg), and mean BP(mmHg) between the CPAP group and the usual care group.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Lin Lee, M.D., PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No